CLINICAL TRIAL: NCT06581861
Title: PREVENT ALL ALS - Longitudinal Biomarker Study for Participants Who Are Genetically at Risk for Amyotrophic Lateral Sclerosis (ALS)
Brief Title: PREVENT ALL ALS Study
Status: Recruiting | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Foundation for the National Institutes of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2024P001131; 1OT2NS136938 (NIH); 1OT2NS136939 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-09-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Biomarker; Observational; at-risk
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ALL ALS Clinical Research Consortium is establishing research to collect a wide range of samples, clinical information and measurements from Amyotrophic Lateral Sclerosis (ALS) symptomatic, ALS gene carriers and control cohorts. This consortium is begin funded by the National Institutes of Health/National Institute of Neurological Disorders and Stroke (NIH/NINDS) and managed by two clinical coordinating centers (CCC) at Barrow Neurological Institute and Massachusetts General Hospital. The clinical sites are distributed across the country, and led by a group of collaborative principal investigators. Once data and samples are collected and harmonized, it will be made available to research community for future research into ALS and related neurological diseases.

PREVENT protocol is specific for asymptomatic participants who are genetically at risk for ALS. The participants will be followed for up to 36 months (3 years), and will include 4 in-person on-site visits once a year and 6 off-site(remote) visits once in 4 months. The study includes collection of medical history, clinical outcomes, and blood samples once in 4 months. Additionally, the participants will complete patient reported outcomes and speech recordings once in 4 months. Participants may also provide optional Cerebrospinal Fluid (CSF) samples.The participants may also opt into a sub-study if they are interested in genetic testing for ALS causative genes. The sub-study will involve a minimum of 3 visits over a course of 2-3 months. This will include a screening/pre-test genetic counseling visit, a return of genetic results and a post-test counseling visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Capable of providing informed consent
3. Willing to follow study procedures
4. First-degree relative of a known carrier of any ALS causative gene1 (regardless of whether ALS or FTD has actually been symptomatic in the family) OR First-degree relative of an individual with ALS and/or FTD in a family with a "compelling family history" of ALS/FTD, regardless of whether genetic testing has occurred in symptomatic family members. A "compelling family history" is defined as a pedigree with at least 2 close relatives who had ALS or FTD, with at least one of those family members having had ALS.
5. Access to a smartphone, computer, or tablet, and internet (need not be in the home - access to a public library or other available computer with internet connection is sufficient)

Exclusion Criteria:

1. Evidence of neurological signs or symptoms concerning for ALS of FTD, at the discretion of the site investigator which will be communicated to the applicant along with referral for appropriate clinical follow-up.
2. Significant cognitive impairment, clinical dementia, or unstable psychiatric illness, including psychosis, active suicidal ideation, suicide attempt, or untreated major depression <= 90 days (about 3 months) of screening, which in the opinion of the Investigator would interfere with the study procedures
3. Clinically significant, unstable medical condition (e.g., cardiovascular instability, systemic infection, untreated thyroid dysfunction, malignant and potentially progressive cancer) that would render the participant unlikely to be able to complete 12 months of follow-up, according to Investigator's judgment

Exclusion Criteria for Participants Undergoing Optional Lumbar Puncture

1. Medically unable to undergo lumbar puncture (LP) as determined by the site investigator (i.e., bleeding disorder, a skin infection at or near the LP site, known or suspected intracranial or intraspinal tumor or other cause of increased intracranial pressure).
2. Allergy to Lidocaine or other local anesthetic agents.
3. Use of anticoagulant medication or antiplatelet medications (aside from aspirin 81 mg) that cannot be safely withheld prior to lumbar puncture.
4. Blood dyscrasia, abnormal bleeding diathesis, or the use of dialysis for renal failure.
5. Current pregnancy based on participant self-report
6. Clinical judgement of the site investigator that the participant would be unable to undergo multiple lumbar punctures.

Inclusion Criteria for Genetic Testing Results Sub-study

1. Age 18 years of age or older
2. Capable of providing informed consent
3. Willing to follow study procedures
4. Currently enrolled in the PREVENT ALS Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 600 participants are planned for this study enrolled. They are aged 18 years or older, and are at risk of developing ALS.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-25 (Estimated)

PRIMARY OUTCOMES:
ALS Symptoms Questionnaire | Baseline, 4, 8, 12,16,20, 24, 28, 32 and 36 months form baseline
  Questions to identify development of symptoms related to ALS

SECONDARY OUTCOMES:
Environmental History | Once at Month 1 from Baseline
  Questionnaires completed by participants that includes questions about non-medical factors that affect health outcomes
Cognitive assessment (ECAS) | at Baseline, 12, 24 and 36 months from baseline
  ECAS is a multi-domain assessment administered by study staff, to evaluate different aspects of cognitive function
Cognitive assessment (CDR-FTLD) | at Baseline, 12, 24 and 36 months from baseline
  CDR-FTLD is a global assessment scale that evaluates severity of impairment across multiple domains in patients with Frontotemporal dementia (FTLD) spectrum disorders.
Hand-Held Dynamometry (HHD) | at Baseline, 12, 24 and 36 months from baseline
  HHD is used as a quantitative measure of muscle strength. This will involve testing of the bilateral deltoid, biceps, triceps, wrist extension, FDI, ADM, APB, hip extension, quadriceps, hamstring, TA and grip strength.
Digital Speech Assessment | at Baseline, and at months 4,8,12,16,20,24,28,32 and 36 months
  Participants will be asked to record voice samples at home once a month using a digital application installed on their device.
Vital Capacity (VC) | at Baseline, 12, 24 and 36 months from baseline
  It is the change in respiratory function over time as measured by Slow Vital Capacity (SVC).

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of California Irvine, Orange, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Nih/Ninds, Bethesda, Maryland
  - Massachusetts General Brigham, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Penn State Health, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- CHALS-CCT, University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico, Puerto Rico